CLINICAL TRIAL: NCT05425537
Title: The Epidemiological Profile of Non-fatal and Fatal Drowning: A Danish Nationwide Registry-based Cohort Study
Brief Title: Drowning in Denmark: A Registry-based Study of Fatal and Non-fatal Drowning From 2016 to 2023
Status: Completed | Type: Observational
Sponsor: Prehospital Center, Region Zealand (Other)
Responsible Party: Principal Investigator, Niklas Breindahl, Medical Doctor, PhD-student, Prehospital Center, Region Zealand
Other Study IDs: DROWN_NONFATAL
Record Dates: First submitted 2022-05-29; First posted 2022-06-21 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Drowning
Keywords: Drowning; Non-fatal; Utstein; Register study; Retrospective; Reigstry-based study
MeSH Terms: conditions — Drowning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fatal drowning: Fatal drowning incident where the patient died because of the drowning process
  Interventions: Other: Drowning incident
- Non-fatal drowning: Non-fatal drowning incident where the patient was drowning and can be ascertained to have been experiencing either mild, moderate, or severe respiratory impairment immediately after the drowning process ended but survived.
  Interventions: Other: Drowning incident

INTERVENTIONS:
Other: Drowning incident — Drowning is defined by the WHO in 2002 as "the process of experiencing respiratory impairment from submersion or immersion in liquid"

SUMMARY:
Using nationwide data from the prehospital electronic health records from 2016 to 2023, this registry-based cohort study aims to establish a nationwide epidemiological profile of non-fatal and fatal drowning patients in Denmark in adherence with the Utstein Style For Drowning (USFD) recommended guidelines for uniform reporting of data from drowning. This includes reporting the annual incidence rates per 100,000 person-years, assessing the associations between predefined prognostic variables and 30-day survival, and reporting the spatial distribution of drowning incidents presented on a map of Denmark.

DETAILED DESCRIPTION:
Purpose

The purpose of this study is to establish a nationwide epidemiological profile of non-fatal and fatal drowning patients in Denmark which can be used to target educational, preventative, rescue, or treatment strategies to reduce the number of fatal and non-fatal drowning incidents in Denmark.

Objectives

The primary objective is to estimate the yearly incidence rates of drowning patients in Denmark treated by the Danish Emergency Medical Services from 2016 to 2023. The secondary objective is to report the associations between predefined prognostic variables and 30-day survival.

Study design

A nationwide registry-based study with data from the Danish Drowning Cohort (extracted from the prehospital electronic health records using syndromic surveillance and extensive manual validation) from 2016 to 2023 with 30-day follow-up.

ELIGIBILITY:
Inclusion criteria:

* The patient must have been experiencing respiratory impairment from submersion or immersion in liquid AND
* The patient must have been in contact with the Danish prehospital emergency medical services.

Exclusion criteria:

- Patients were excluded if the incident involved submersion or immersion with aspiration, but the patient did not experience respiratory impairment. For example, if the patient was rescued from the water without signs of respiratory impairment, or if the respondent reported "a few coughs" or "voluntary cough".

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All drowning patients who have been treated by the Danish prehospital emergency medical services in the period from 2016-2023.
Sampling Method: Probability Sample
Enrollment: 1664 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Annual drowning incidence rates per 100,000 person-years from 2016-2023 | Counts of fatal and non-fatal drowning incidents will be obtained between 2016-2023.
  The primary objective is to estimate the annual incidence of fatal and non-fatal drowning patients in Denmark treated by the prehospital emergency medical services from 2016 to 2023 and will be reported as the annual number of cases per 100,000 person-years.
30-day survival following drowning incidents in Denmark from 2016-2023 | 30-day follow-up after the drowning incident
  The primary outcome is 30-day survival (alive/dead).

SECONDARY OUTCOMES:
Association between prognostic variables and 30-day survival | From 2016-2023
  This outcome will explore predefined prognostic variables associated with 30-day survival after a drowning incident. The following risk factors will be analysed using multivariable logistic regression models and presented as odds ratios (ORs) with 95% confidence intervals (CIs): witnessed status, sex, age, OHCA, submersion duration, season, location.
Map of fatal and non-fatal drowning incidents in Denmark from 2016-2023 | From 2016-2023
  Showing a map of geographical localization of drowning in Denmark in the study period indicating 30-day mortality and survival

CONTACTS AND LOCATIONS:
Overall Officials: Niklas Breindahl, MD, PhD, Principal Investigator — Prehospital Center, Region Zealand
Locations (1):
- Prehospital Center, Næstved, Region Sjælland, Denmark

REFERENCES:
- [Background] Weiss J; American Academy of Pediatrics Committee on Injury, Violence, and Poison Prevention. Prevention of drowning. Pediatrics. 2010 Jul;126(1):e253-62. doi: 10.1542/peds.2010-1265. Epub 2010 May 24. PMID 20498167
- [Background] Schmidt AC, Sempsrott JR, Szpilman D, Queiroga AC, Davison MS, Zeigler RJ, McAlister SJ. The use of non-uniform drowning terminology: a follow-up study. Scand J Trauma Resusc Emerg Med. 2017 Jul 17;25(1):72. doi: 10.1186/s13049-017-0405-x. PMID 28716063
- [Background] Papa L, Hoelle R, Idris A. Systematic review of definitions for drowning incidents. Resuscitation. 2005 Jun;65(3):255-64. doi: 10.1016/j.resuscitation.2004.11.030. PMID 15919561
- [Background] Lu TH, Lunetta P, Walker S. Quality of cause-of-death reporting using ICD-10 drowning codes: a descriptive study of 69 countries. BMC Med Res Methodol. 2010 Apr 8;10:30. doi: 10.1186/1471-2288-10-30. PMID 20374660
- [Background] Steensberg J. Epidemiology of accidental drowning in Denmark 1989-1993. Accid Anal Prev. 1998 Nov;30(6):755-62. doi: 10.1016/s0001-4575(98)00028-1. PMID 9805518
- [Background] Mackie IJ. Patterns of drowning in Australia, 1992-1997. Med J Aust. 1999 Dec 6-20;171(11-12):587-90. doi: 10.5694/j.1326-5377.1999.tb123808.x. PMID 10721338
- [Background] Truhlar A, Deakin CD, Soar J, Khalifa GE, Alfonzo A, Bierens JJ, Brattebo G, Brugger H, Dunning J, Hunyadi-Anticevic S, Koster RW, Lockey DJ, Lott C, Paal P, Perkins GD, Sandroni C, Thies KC, Zideman DA, Nolan JP; Cardiac arrest in special circumstances section Collaborators. European Resuscitation Council Guidelines for Resuscitation 2015: Section 4. Cardiac arrest in special circumstances. Resuscitation. 2015 Oct;95:148-201. doi: 10.1016/j.resuscitation.2015.07.017. Epub 2015 Oct 15. No abstract available. PMID 26477412
- [Background] Venema AM, Groothoff JW, Bierens JJ. The role of bystanders during rescue and resuscitation of drowning victims. Resuscitation. 2010 Apr;81(4):434-9. doi: 10.1016/j.resuscitation.2010.01.005. Epub 2010 Feb 10. PMID 20149515
- [Background] Idris AH, Berg RA, Bierens J, Bossaert L, Branche CM, Gabrielli A, Graves SA, Handley AJ, Hoelle R, Morley PT, Papa L, Pepe PE, Quan L, Szpilman D, Wigginton JG, Modell JH; American Heart Association. Recommended guidelines for uniform reporting of data from drowning: the "Utstein style". Circulation. 2003 Nov 18;108(20):2565-74. doi: 10.1161/01.CIR.0000099581.70012.68. No abstract available. PMID 14623794